CLINICAL TRIAL: NCT02809703
Title: Assessment of the Long Term Quality of Life Following Veno-venous and Veno-arterial Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: Quality of Life Following ECMO
Status: Withdrawn | Type: Observational
Why Stopped: PI departed study site. Study closed.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00070210
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Extracorporeal Membrane Oxygenation; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey Questions — Subjects will receive surveys via direct mail. They will be given the opportunity to opt in to receive a phone call regarding quality of life.

SUMMARY:
The objective of the study is to determine the quality of life of patients in the years following treatment with extracorporeal membrane oxygenation (ECMO). The study population will include all adults treated with any configuration of ECMO at Duke University Medical Center during the period of Jan 1, 2009 and Dec 31, 2015. Patient's will be contacted by direct mail, in conjunction with a surgeon who performed their ECMO procedure or managed them while on ECMO, and asked to complete a validated survey (WHOQOL-Bref) which assesses quality of life. In addition, patients will be asked to opt-in to participate in a phone survey in which they can give a narrative about their ICU experience and answer specific questions regarding long-term comorbidities. Data will be stored in a secure online server which is HIPAA compliant and analyzed by the department of anesthesiology statistical support services. De-identified data will be shared with the WHO as specified in their usage agreement.

ELIGIBILITY:
Inclusion Criteria:

* VA or VV ECMO performed during retrospective study period

Exclusion Criteria:

* Pediatric

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent VV or VA ECMO at Duke.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Quality of Life as Assessed by the WHOQOL-BREF. | 6 months to 5 years post ECMO procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States